CLINICAL TRIAL: NCT01903486
Title: A Pilot Study Assessing the Efficacy of Steroids in the Treatment of Achalasia
Brief Title: Assessing the Efficacy of Steroid Treatment of Achalasia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit participants.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karthik Ravi, M.D., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-009825
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Achalasia
Keywords: Trouble swallowing; dysphagia; disorder of the esophagus
MeSH Terms: conditions — Esophageal Achalasia; Deglutition Disorders | interventions — Prednisone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prednisone (Other): Prednisone (study medication) at a dose of 40mg for 1 week, then 30mg for 1 week, then 20mg for 1 week, then 10mg for 1 week, and then stop the medication.
  Interventions: Drug: Apo-Prednisone Cordorol, Detasone - Prednisone

INTERVENTIONS:
Drug: Apo-Prednisone Cordorol, Detasone - Prednisone — Oral prednisone (study medication) at a dose of 40mg for 1 week, then 30mg for 1 week, then 20mg for 1 week, then 10mg for 1 week, and then stop the medication.
  Other Names: Prednisone; Anti-inflamatory; Corticosteroid

SUMMARY:
Would systemic steroids be an effective treatment in early variants of achalasia?

ELIGIBILITY:
Inclusion criteria:

* Adults ages 18-90 with a diagnosis of achalasia confirmed by findings on esophageal manometry and barium esophagogram will be eligible for the study.
* Eckardt score6 greater or equal to 6 or 2 or greater for dysphagia and/or regurgitation
* Symptoms less than 2 years

Exclusion criteria:

* Medical conditions such as severe heart or lung disease that preclude safe performance of endoscopy and injection;
* Greater than mild esophageal dilation
* Type 1 achalasia as defined by the Chicago classification scheme7 and/or esophageal diameter > 3cm;
* Prior treatment for achalasia
* Use of medications that might affect LES pressure such as anticholinergics or calcium channel antagonists
* Symptom duration greater than 2 years
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy
* Disorders which predispose to unreliable responses such as Schizophrenia, Alzheimer's disease or significant memory loss
* Pregnant and lactating females will be excluded as steroids are not thought safe for the fetus.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
the proportion of patients with an Eckhart score ≥ 6 at 1 month | Baseline to 1 month

SECONDARY OUTCOMES:
proportion of patients with symptomatic improvement (Eckardt sore 6 or greater) | baseline to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ravi, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials